CLINICAL TRIAL: NCT05911737
Title: Ocular Parameters Assessment With a Deep Neural Network in Patients With Sleep Apnea
Brief Title: Ocular Parameters in Patients With Sleep Apnea
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Professor (Associate) of Democritus University of Thrace, Democritus University of Thrace
Other Study IDs: ES2/Th35/27-02-2020
Record Dates: First submitted 2023-06-10; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Sleep Apnea Syndrome, Obstructive; Drowsiness; Blinking; Concentration Ability Impaired; Pupil Diameter
Keywords: Reading Time; Fixation; Saccadic movements; Eyelid margin distance
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleepiness | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients diagnosed with Obstructive Sleep Apnea: Patients diagnosed with Obstructive Sleep Apnea
  Interventions: Behavioral: Short video and Questionnaire
- Patients not diagnosed with Obstructive Sleep Apnea: Patients not diagnosed with Obstructive Sleep Apnea
  Interventions: Behavioral: Short video and Questionnaire

INTERVENTIONS:
Behavioral: Short video and Questionnaire — A 10-minute video in a foreign language (not English or Greek) with greek subtitles will be presented and a questionnaire will follow to assess the level of concentration during the video

SUMMARY:
The aim of this study is to assess the ocular parameters of drowsiness in patients with diagnosed Obstructive Sleep Apnea Syndrome through objective methods of ocular imaging and subjective evaluation methods (questionnaire)

DETAILED DESCRIPTION:
This is a single-center prospective comparative observational study. One hundred patients with drowsiness that will be examined in the Sleep Clinic of Alexandroupolis University Hospital, aged between18-70 years old, with Distance Uncorrected Visual Acuity ≥ (dUVA): 5/10 will be recruited. They will be separated into two groups, one consisting of patients with diagnosed Obstructive Sleep Apnea and one without this diagnosis, according to the Epworth Sleepiness Scale - ESS, which is a valid tool for quantifying daily sleepiness. A 10-minute video in a foreign language (not English or Greek) with greek subtitles will be presented to them and a questionnaire will follow to assess the level of concentration during the video (the subtitles are crucial to understanding the video's plot). The video will be displayed in a 11.6" screen with resolution of 1920x1080 pixels, at 70 cm patient-to-screen distance. The patients' eyes will be recorded during the video with a Raspberry Pi Camera Module IR-CUT v2 (5MP,1080p) with 2 IR LED lights, connected to a Raspberry Pi 3 model v1.2, operating at the original resolution of 1080×1920, at 20 cm patient-to-camera distance and an algorithm will be developed to analyze the following parameters: 1. The complete and incomplete blinks defined by the "length of palpebral fissure-to-iris diameter" ratio, 3. Length of palpebral fissure of both eyes.

ELIGIBILITY:
Inclusion Criteria:

* patients with obstructive sleep apnea and controls, aged 18-70 years old, with distance uncorrected visual acuity (dUVA) ≥ 5/10.

Exclusion Criteria:

* (dUVA) <5/10,
* intraocular pressure lowering medications
* former corneal or fundus disease
* neurological or psychiatric conditions
* mental disability
* difficulty reading

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with obstructive sleep apnea and controls (not diagnosed with οbstructive sleep apnea)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Total number of blinks during the 10-minute video | 1 week
  The total number of blinks during the 10-minute video. Complete blinks are defined by the "length of palpebral fissure-to-iris diameter" ratio.
Total number of complete blinks during the 10-minute video | 1 week
  The total number of complete blinks during the 10-minute video. Complete blinks are defined by the "length of palpebral fissure-to-iris diameter" ratio.
Total number of incomplete blinks during the 10-minute video | 1 week
  The total number of incomplete blinks during the 10-minute video. Incomplete blinks are defined by the "length of palpebral fissure-to-iris diameter" ratio.
Number of total blinks for each minute | 1 week
  Number of total blinks for each minute of the 10-minute video
Number of complete blinks for each minute | 1 week
  Number of complete blinks for each minute of the 10-minute video
Number of incomplete blinks for each minute | 1 week
  Number of incomplete blinks per minute for each minute of the 10-minute video
Total blinks per minute | 1 week
  Total blinks per minute during the 10-minute video
Complete blinks per minute | 1 week
  Complete blinks per minute during the 10-minute video
Incomplete blinks per minute | 1 week
  Incomplete blinks per minute during the 10-minute video
Length of palpebral fissure of both eyes | 1 week
  The distance between the upper eyelid margin and the lower eyelid margin (ie. the vertical dimension of the palpebral fissure) for each frame

SECONDARY OUTCOMES:
Fixations to the area of interest | 1 week
  Number of fixations to the area of interest (subtitles)
Fixation duration | 1 week
  Mean fixation duration (duration of fixation per video per participant)
Reading time | 1 week
  The absolute reading time (the sum of the duration of all fixations and saccadic movements in the area of focus starting from the first fixation)
Participant's dedication time to the area of focus | 1 week
  The percentage of time that each participant dedicates to the area of focus depending on the time of subtitle exposure (eg. subtitle reading time/overall subtitle exposure= 2500 msec/3000 msec=83%)
Rereadings | 1 week
  Rereadings: the number of fixations/seccadic movements to the area of focus after the first reading (indicating of subtitlte interpretation difficulty or extended subtitle exposure time).

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, PhD, Study Chair — Democritus University of Thrace
Locations (1):
- Democritus University of Thrace, Alexandroupoli, Evros, Greece